CLINICAL TRIAL: NCT06405529
Title: Rehabilitation of Patients Submitted to Mechanical Ventilation, From the ICU to the Post-hospital Phase: Blinded Randomized Controlled Clinical Trial, With Economic and Multicenter Evaluation
Brief Title: Rehabilitation of Patients From the ICU to the Post-hospital Phase
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, Professor, PhD Physiotherapist, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: USP-2024
Record Dates: First submitted 2024-01-07; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Early Mobilization; Physiotherapy; Rehabilitation
Keywords: Mechanical ventilation; Physiotherapy; Respiratory function; Functional capacity; Rehabilitation; Cost-effectiveness
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): During hospitalization in the ICU and ward, this group will perform a maximum of 10 minutes of exercises of the casual care per day.
- Intervention Group (Experimental): During hospitalization in the ICU and ward, this group will perform 30 to 60 minutes of exercises per day, according to the IMS scale and the intensive mobilization protocol.
  Interventions: Other: Early and intensive mobilization protocol at the ICU and Rehabilitation post-hospital discharge
- Guidance Group (No Intervention): After hospital discharge, this group will not participate in any supervised exercise session, they will only be instructed by the therapists and receive the exercise booklet from the Rehabilitation Center.
- Rehabilitation Group (Experimental): After hospital discharge, this group will participate in a supervised exercise program twice a week for 8 weeks at the Rehabilitation Center.
  Interventions: Other: Early and intensive mobilization protocol at the ICU and Rehabilitation post-hospital discharge

INTERVENTIONS:
Other: Early and intensive mobilization protocol at the ICU and Rehabilitation post-hospital discharge — During hospitalization in the ICU and ward, you will perform 30 to 60 minutes of exercises per day, according to the IMS scale.
  After hospital discharge, participation in a supervised exercise program twice a week for 8 weeks at the Rehabilitation Center - CER of the Hospital das Clínicas of the Faculty of Medicine of Ribeirão Preto.
  Arms: Intervention Group; Rehabilitation Group

SUMMARY:
Introduction: Advances in knowledge have contributed to the increase in the number of patients who survive prolonged hospitalization in an Intensive Care Unit (ICU), and, among them, critically ill patients who develop acute respiratory failure and need for mechanical ventilation. These individuals have their mobility restricted to bed, and may suffer from pulmonary and systemic complications, such as ICU-Acquired Muscle Weakness, which increases the chances of resulting in reduced functional capacity or death. Early mobilization in the ICU has demonstrated benefits, but still with a low level of evidence. However, the type and intensity of exercise still need to be better defined, and previous protocols did not offer continuous monitoring from the ICU to the ward and subsequent outpatient rehabilitation for these patients, which is considered a limitation in some studies.

Objective: To investigate the effects of an early and intensive hospital mobilization and post-hospital rehabilitation program on indicators of functionality, inflammation, cost-effectiveness, and mortality in critically ill patients undergoing invasive mechanical ventilation.

Methods: This is a Blind Randomized Controlled Clinical Trial that will be conducted in the ICUs of the Hospital das Clinicas and the Emergency Unit of the Faculty of Medicine of Ribeirao Preto of the University of São Paulo. Patients of both sexes over 21 years of age who have been under invasive mechanical ventilation for at least 24 hours will be recruited. Patients will be randomized into the Intervention Group (IG), with 30 to 60 minutes of exercise per day, and the Control Group (CG), with 10 minutes of exercise per day, both with the same protocol and based on the ICU Mobility Scale - IMS, with continuity in the ward. After hospital discharge, participants will be allocated to the Guidance Group (GIor and GCor) and the Outpatient Rehabilitation Group (GIreab and GCreab), with functional exercise capacity as the main outcome, assessed by the six-minute walk test (6MWT). Volunteers will be monitored one, three, and six months after hospital discharge. The sample calculation was based on the results of the 6MWT , with a power of 80% for the assessments carried out at the proposing institution (n=206), and with a power of 90% for the multicenter project (n=275), considering a sample loss of 30%. The following will be evaluated: clinical parameters, severity indexes, functionality, lung function and mechanics, functional exercise capacity, mortality, inflammatory markers, energy expenditure, activities of daily living, quality of life, muscle assessment, adherence, barriers and facilitators and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age greater than or equal to 21 years
* Be on invasive mechanical ventilation (IMV) for at least 48 hours
* Sufficient cardiovascular stability for mobilization

  1. Absence of bradyarrhythmia (< 50 bpm);
  2. Heart rate ≥ 150 bpm;
  3. Most recent lactate measurement ≤ 4.0mmol/L;
  4. Combined adrenaline/noradrenaline infusion rate ≤ 0.2mcg/Kg/min, OR if the adrenaline/noradrenaline infusion was increased by more than 25% in the last 6 hours;
  5. Cardiac index ≥ 2.0L/min/m2; when evaluated
* Respiratory stability sufficient for mobilization f) Respiratory rate ≤ 45rpm; g) FiO2 ≤ 0.6; h) PEEP ≤ 16 cmH2O; i) No need for NO (nitric oxide), prone position, neuromuscular blocker, ECMO (extracorporeal membrane oxygenation) or HFOV (high frequency ventilation).

Exclusion Criteria:

* Dependent for ADLs in the month prior to ICU admission;
* Diagnosed cognitive deficit;
* Diagnosis OR suspicion of acute primary brain disease (TBI, stroke);
* Diagnosis OR suspected spinal cord injury OR other neuromuscular disease that may result in prolonged or permanent muscle weakness (except muscle weakness acquired in the ICU);
* Need OR instructions to remain in bed OR not to bear weight on the lower limbs bilaterally;
* Life expectancy of less than 180 days due to acute or chronic clinical conditions;
* Death considered inevitable due to current clinical condition or if the patient/clinical guardian is not committed to complete active treatment (e.g. brain death);
* Inability to communicate in Portuguese;
* Readmission to the ICU of the same hospital service;
* Pregnant women;
* Patients with a permanent pacemaker.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | Through study completion, an average of 5 year
  Assessed by the 6-minute walk test

SECONDARY OUTCOMES:
Clinical parameters | Through study completion, an average of 5 year
  Hemodynamic data will be evaluated beafore and after the mobilization protocol
Clinical parameters | Through study completion, an average of 5 year
  Level of sedation evaluated by the Richmond Agitation-Sedation Scale (RASS). The scale ranges from -4 to +5, from the highest level of agitation to coma.
Clinical parameters | Through study completion, an average of 5 year
  Length of stay in the ICU (tICU) and Length of hospital stay (LoS)
Clinical parameters | Through study completion, an average of 5 year
  Time on mechanical ventilation (tMV)
Severity indexes | Through study completion, an average of 5 year
  Acute Physiologic and Chronic Health Evaluation II Score (APACHE II). This tool assesses the severity of the disease and mortality of patients admitted to the ICU, consisting of 12 variables that include: age, past medical history, as well as clinical and physiological indices.
Severity indexes | Through study completion, an average of 5 year
  Sequential Organ Failure Assessment Score (SOFA Score). This tool calculates both the number and severity of organic dysfunction in six organic systems (respiratory, coagulation, hepatic, cardiovascular, renal and neurological).
Pulmonary function | Through study completion, an average of 5 year
  Spirometry will be used as a tool to assess the lung function. The test will be performed by every volunteer and the measurement will be done by guidelines of the Brazilian Society of Pulmonology and Phthisiology for lung function tests.
Pulmonary function | Through study completion, an average of 5 year
  Impulse oscillometry system (IOS). This test will be perfomed to evaluate the resistance of the respiratory system in accordance with that proposed by Oosteveen (2003).
Pulmonary function | Through study completion, an average of 5 year
  Diffusing capacity of the lungs for carbon monoxide (DLCO). This is a pulmonary function test used to assess the lungs' ability to transfer gas from inspired air to the bloodstream. Normal severity slassification is up to 75% of the predicted value.
Pulmonary function | Through study completion, an average of 5 year
  Computed tomography (CT). The high-resolution CT technique with low dose of radiation will be used, without the administration of iodinated contrast medium, scanning the entire chest in the caudocranial direction, with volumetric acquisition of 1 mm in thickness during complete inspiration. Quantitative analysis of HRCT images will be performed using the scientific program Yacta version 2.8 (Heussel et al., 2009).
Mortality | Through study completion, an average of 5 year
Cost-effectiveness | 12 months after study completion
  Economic evaluation - Patient and Institution costs

IPD SHARING:
Plan to Share IPD: Yes